CLINICAL TRIAL: NCT00006994
Title: S9908, A Double-Blind, Placebo-Controlled Trial To Study The Efficacy And Safety Of L-Glutamine (In AES0014 Delivery Vehicle) Upon Radiation Therapy-Induced Oral Mucositis In Head and Neck Cancer Patients, Phase III
Brief Title: S9908: Glutamine in Treating Mucositis Caused by Radiation Therapy in Patients With Newly Diagnosed Cancer of the Mouth or Throat
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn due to drug availability and funding
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000068353; S9908 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Cancer-related Problem/Condition; Head and Neck Cancer; Pain
Keywords: oral complications of radiation therapy; pain; radiation toxicity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Pain; Radiation Injuries; Squamous Cell Carcinoma of Head and Neck | interventions — Glutamine; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-glutamine in suspension + radiation (Active Comparator): 20 cc three times daily for 60 days plus radiation therapy.
  Interventions: Dietary Supplement: glutamine; Radiation: radiation therapy
- Placebo in suspension + radiation (Placebo Comparator): 20 cc three times daily for 60 days plus radiation therapy.
  Interventions: Radiation: radiation therapy; Drug: l-glutamine placebo

INTERVENTIONS:
Dietary Supplement: glutamine — 20 cc three times daily for 60 days
  Other Names: l-glutamine; NSC-143503
  Arms: L-glutamine in suspension + radiation
Radiation: radiation therapy — Per institutional standard; minimum of 6,000 cGy with a daily dose of 180-200 cGy.
Drug: l-glutamine placebo — 20 cc three times daily for 60 days
  Other Names: NSC-143503
  Arms: Placebo in suspension + radiation

SUMMARY:
RATIONALE: Glutamine may be effective in decreasing side effects, such as inflammation of the mouth and throat, caused by radiation therapy. The effectiveness of glutamine for mucositis is not yet known.

PURPOSE: Randomized phase III trial to determine the effectiveness of glutamine in treating patients who develop mucositis following radiation therapy for newly diagnosed cancer of the mouth or throat.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of L-glutamine vs placebo, in terms of maximum mucositis toxic effects and worst reported mouth pain during and after high-dose radiotherapy, in patients with newly diagnosed, previously untreated squamous cell cancer of the oral cavity or oropharynx.
* Compare the duration of severe mucositis in patients treated with these regimens.
* Compare the radiotherapy delay in patients treated with these regimens.
* Compare weight loss in patients treated with these regimens.
* Compare the toxic effects of these two regimens in these patients.
* Compare patient-reported mouth pain success rate in patients treated with these regimens.
* Determine the compliance of patients treated with this drug regimen.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to concurrent cisplatin or carboplatin (yes vs no), concurrent fluorouracil (yes vs no), and presence of feeding tube (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning 4 to 7 days prior to radiotherapy, patients receive oral L-glutamine 3 times daily for 60-80 days. Patients receive concurrent high-dose radiotherapy for approximately 6 weeks.
* Arm II: Patients receive oral placebo and high-dose radiotherapy as in arm I. In both arms, treatment continues in the absence of unacceptable toxicity.

Patients are followed for 2 weeks.

PROJECTED ACCRUAL: A total of 158 patients (79 per treatment arm) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed, previously untreated squamous cell cancer of the oral cavity or oropharynx (T1-T4, any N, M0)
* Must be scheduled to receive high-dose radiotherapy
* Not concurrently receiving or planning to receive treatment on any other Southwest Oncology Group protocol

PATIENT CHARACTERISTICS:

Age:

* 18 to 90

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage I or II cancer currently in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* Concurrent cisplatin, carboplatin, or fluorouracil allowed
* No other concurrent chemotherapy during study and for at least 3 weeks after study radiotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Other:

* No concurrent amifostine during and for 2 weeks after study radiotherapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-11; Primary Completion 2005-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of L-glutamine for mucositis | 2 weeks after end of radiation treatment
  Evaluate effectiveness of L-glutamine as compared to placebo in terms of: maximum toxicity grade during radiation treatment, mucositis toxicity grade 2 weeks after the end of radiation treatment, and patient reported worst mouth pain two weeks after the end of radiation treatment.

SECONDARY OUTCOMES:
Duration of severe mucositis, radiation treatment delay, and weight loss | 2 weeks after radiation treatment
Toxicities | within 2 weeks after radiation treatment
Compare patient reported mouth pain "success" rate at the end of radiation treatment | 2 weeks after end of radiation treatment
Compliance (dose taken) in patients treated with L-glutamine when given with radiation treatment | 2 weeks after end of radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: V. S. Klimberg, MD, Study Chair — University of Arkansas
Locations (107):
- United States (106):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Hospital Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Veterans Affairs Medical Center - Salisbury, Salisbury, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Danville Radiation Therapy Center, Memphis, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada